CLINICAL TRIAL: NCT04455438
Title: Phase I Trial Evaluating Stereotactic Body Radiotherapy (SBRT) Dose Escalation for Reirradiation of Inoperable Lung Lesions
Brief Title: SBRT Dose Escalation for Reirradiation of Inoperable Lung Lesions
Acronym: STRILL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2525
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Non Small Cell Lung Cancer; Lung Metastases
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: The study is designed to determine the Maximum Tolerated Dose (MTD) that could be safely delivered in the lung reirradiation setting. The MTD was defined as the highest dose level in which a proportion of 1 out of 5 or fewer patients experienced DLT. Due to the late onset nature of DLT, in order to allow for continuous accrual without sacrificing patient safety or the accuracy of identifying the MTD, the Time-To-Event Bayesian Optimal Interval (TITE-BOIN) design will be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SBRT Level 1 (Experimental): The starting dose level will be SBRT 30 Gy in 5 fractions (level 1 or L1).
  Interventions: Radiation: SBRT dose escalation
- SBRT Level 2 (Experimental): If the starting dose is tolerated in the first 5 patients, the next dose will be SBRT 40 Gy in 5 fractions (level 2 or L2)
  Interventions: Radiation: SBRT dose escalation
- SBRT Level 3 (Experimental): If the second dose is tolerated in the next 5 patients, the next dose will be SBRT 50 Gy in 5 fractions (level 3 or L3)
  Interventions: Radiation: SBRT dose escalation

INTERVENTIONS:
Radiation: SBRT dose escalation — Re-Stereotactic Body Radiation Therapy (SBRT) with increasing dose levels, from 30 Gy in 5 fractions to 50 Gy in 5 fractions.

SUMMARY:
Prospective phase I study to evaluate the maximum tolerated dose (MTD) of SBRT for thoracic re-irradiation. Dose limiting toxicity will be pneumonitis ≥ G3. The potential advantage of the dose escalation planned in this study is the delivery of an ablative dose to radically treat patients with inoperable local relapse, without unacceptable toxicity.

DETAILED DESCRIPTION:
Radical dose radiotherapy (RT) is frequently used in thoracic malignancies, both for early stage primary non-small cell lung cancer (NSCLC) and for secondary lesions from other primary tumors, particularly in the setting of oligometastatic patients. Although development of distant metastases is the predominant pattern of failure after treatment with radical RT, isolated local recurrences, defined as a tumor recurrence overlapping the 50% isodose field, are still observed and are becoming more and more frequent along with the prolongation of life expectancy in cancer patients. Salvage options for isolated post-radiation local failures are limited, with surgery or retreatment with radiotherapy as potential modalities.

While salvage surgical resection after previous thoracic irradiation has shown encouraging results, most patients experiencing post-radiation local relapse are not surgical candidates. Therefore, reirradiation may be the only viable salvage option for many patients. Retreatment with CFRT has been reported for locoregional failures, with generally-poor outcomes. Although, salvage SBRT after initial CFRT has been described in select small series of heterogeneous patient groups ranging from early stage to locally-advanced and metastatic, few data exist to guide us on the role of reirradiation with SBRT for isolated recurrences after initial SBRT for early-stage NSCLC. Due to the heterogeneity and the low numerosity of these experiences, important questions regarding the safety and efficacy in this setting are still largely unanswered. Particularly, the possibility of delivering a second course of ablative dose RT (BED ≥ 100 Gy) is almost unexplored.

Based on this background, we designed a prospective phase I study to evaluate the maximum tolerated dose (MTD) of SBRT for thoracic re-irradiation. Dose limiting toxicity will be pneumonitis ≥ G3. The potential advantage of the dose escalation planned in this study is the delivery of an ablative dose to radically treat patients with inoperable local relapse, without unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Inoperable primary non-small cell lung cancer or other metastatic primaries with lung metastases, already treated with radical dose RT;
* Peripheral lesion (> 2 cm from trachea-bronchial tree);
* Inoperable local recurrence (defined as a tumor recurrence overlapping the 50% isodose field) confirmed by documented radiographic findings and/or pathological biopsies within the thoracic area;
* Patients had previously received curative intent RT of more than 50 Gy for conventionally fractionated RT or a biologically equivalent dose of more than 75 Gy for SBRT;
* No active distant metastasis or controlled distant metastasis at the time of re-irradiation

Exclusion Criteria:

* Central or ultra-central lesion(s);
* Incapability of understanding and signing informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-05-28 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
MTD | 5 years
  maximal tolerated dose (MTD) of SBRT for thoracic re-irradiation

SECONDARY OUTCOMES:
Other toxicities | 5 years
  To evaluate acute and late toxicities other than dose limiting toxicity
Overall survival | 5 years
  To evaluate overall survival of patients undergoing thoracic re-irradiation.
Local control | 5 years
  To evaluate local control of patients undergoing thoracic re-irradiation.
PFS | 5 years
  To evaluate progression free survival of patients undergoing thoracic re-irradiation.

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No